CLINICAL TRIAL: NCT01146262
Title: Vaccination by Leukemic Apoptotic Corpse Autologous Pulsed Dendritic Cells for AML Patients in First or Second CR
Brief Title: Vaccination by Leukemic Apoptotic Corpse Autologous Pulsed Dendritic Cells for Acute Myelogenous Leukemia (AML) Patients in First or Second Complete Remission (CR)(CD laM)
Acronym: CD lam
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/05/10-L
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Antitumoral immune response after autologous dendritic cells vaccination
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cell therapy product — Patients receive for up to 5 doses of apoptotic corpse pulsed dendritic cells after CR1 ou CR2 documentation (9/10 subcutaneously and 1/10 intradermally) every week, except the last injection performed at 2 weeks from the 4th injection.
Procedure: injection of the cell therapy product — Cytapheresis D0: 1st injection of the cell therapy product, J7 2nd injection of the cell therapy product, J14 third injection of the cell therapy product,J17 cutaneous biopsies, J21 fourth injection of the cell therapy product, J35 fifth injection of the cell therapy product

SUMMARY:
Dendritic cells vaccinations are increasingly used in order to develop antitumoral immune response. This will be a Phase 2 trial using autologous dendritic cells pulsed with leukemic apoptotic corpse in acute myelogenous leukemia (AML) patients in first or second Complete remission (CR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Informed consent signed
* Serology HIV, hepatitis B, hepatitis C, HTLV 1 and 2 and Syphilis always negative (new achievement tests)
* Performance Statute <=2
* Must not be eligible for allogeneic transplantation
* No progressive disease
* Bone marrow and/or peripheral blasts >50% before chemotherapyBlasts >=2.4 10*8 (collected prior to chemotherapy) available No contraindication to cytapheresis
* AML in CR2, except M3-AML
* Patients with refractory AML after induction treatment and a patient eligible for salvage treatment may allow the production of a first complete remission.
* Patient with newly diagnosed AML with unfavorable cytogenetics and for whom (which) a course of intensive induction and consolidation treatment for outpatients are possible
* Patient with newly diagnosed AML with a non-adverse cytogenetics AND either refused to participate in the protocol GOELAMS LAMS-2007, against the exclusion criteria, indicating participation in the protocol GOELAMS LAMS-2007 and for whom (which) a course of induction and intensive out patient treatment for consolidation are possible
* Absence of donor HLA-compatible family or non-family and absence of placental blood available for performing an allograft.

Exclusion Criteria

* Patients who, for reasons psychological, social or geographical boundaries, could be monitored during the study
* No infections or visceral (cardiac, lung, brain, ...) serious uncontrolled
* History of positive allogeneic bone marrow or solid organ transplantation.
* Previous history of autoimmune disease other than vitiligo
* History of other cancer, except cervical carcinoma in situ or basal cell carcinoma of the skin unless deemed cured for over 5 years.
* Inability to collect at the diagnosis of relapsed AML, enough leukemic cells (> 2.4 x108)
* Inability to collect during remission, a sufficient number of monocytes in two leukapheresis maximum
* Failure to obtain a maturation of monocytes
* Patient with AML 3
* Patient may receive an allogeneic hematopoietic stem cell
* No treatment related to treatment of molecules in preclinical development underway or completed MA within the last 4 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 6 weeks
  Primary objective: assess the tolerability of autologous apoptotic corps pulsed dendritic cells vaccine in acute myelogenous leukemia patients in first or second Complete remission. (CR2)

SECONDARY OUTCOMES:
immune response | Day 14
Complete remission | 18 months
Survival | 18 months after injection
  Overall survival (from the documentation of the second RC)

OTHER OUTCOMES:
genomic analysis of dendritic cells | D7

CONTACTS AND LOCATIONS:
Locations (1):
- Cellule de Promotion de la recherche clinique, Nantes, France

REFERENCES:
- [Derived] Chevallier P, Saiagh S, Dehame V, Guillaume T, Peterlin P, Bercegeay S, Le Bris Y, Bossard C, Gauvrit I, Dreno B, Juge-Morineau N, Bene MC, Gregoire M. A phase I/II feasibility vaccine study by autologous leukemic apoptotic corpse-pulsed dendritic cells for elderly AML patients. Hum Vaccin Immunother. 2021 Oct 3;17(10):3511-3514. doi: 10.1080/21645515.2021.1943991. Epub 2021 Jun 21. PMID 34152898